CLINICAL TRIAL: NCT02688556
Title: A Randomized, Multicenter, Double-Masked, Vehicle-Controlled Study of the Safety and Efficacy of OTX-101 in the Treatment of Keratoconjunctivitis Sicca
Brief Title: Phase 3 Study of OTX-101 in the Treatment of Keratoconjunctivitis Sicca
Acronym: Emerald
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OTX-101-2016-001
Record Dates: First submitted 2016-02-13; First posted 2016-02-23 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2021-11

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: KCS; dry eye; cyclosporine
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OTX-101 0.09% (Experimental): 0.09% cyclosporine nanomicellar ophthalmic solution
  Interventions: Drug: cyclosporine
- Vehicle (Placebo Comparator): vehicle of OTX-101
  Interventions: Drug: vehicle of OTX-101

INTERVENTIONS:
Drug: cyclosporine
  Other Names: Seciera
  Arms: OTX-101 0.09%
Drug: vehicle of OTX-101
  Arms: Vehicle

SUMMARY:
This is a randomized, double-masked, vehicle-controlled study of the safety and efficacy of OTX-101 (0.09% cyclosporine nanomicellar solution) in the treatment of keratoconjunctivitis sicca to be conducted at approximately 50 sites.

ELIGIBILITY:
Inclusion Criteria:

* History of dry eye syndrome (KCS) for a period of at least 6 months
* Clinical diagnosis of bilateral KCS
* Lissamine green conjunctival staining sum score of ≥ 3 to ≤ 9 out of a total possible score of 12 (scoring excludes superior zones 2 and 4) in the same eye at both the Screening and Baseline Visits.
* Global symptom score (SANDE) ≥ 40 mm at both the Screening and Baseline Visits
* Corrected Snellen visual acuity (VA) of better than 20/200 in each eye.

Exclusion Criteria:

* Use of cyclosporine ophthalmic emulsion 0.05% (Restasis®) within 3 months prior to the Screening Visit.
* Previous treatment failure (lack of efficacy) with cyclosporine ophthalmic emulsion 0.05% (Restasis).
* Diagnosis of Sjögren's disease ˃ 5 years prior to the Screening Visit.
* Clinical diagnosis or any history of seasonal and/or perennial allergic conjunctivitis.
* Use of systemic or topical medications within 7 days prior to the Screening Visit or during the study period that are known to cause dry eye.
* Use of any topical ophthalmic medications, prescription (including anti-glaucoma medications) or over the counter (including artificial tears), other than the assigned study medication during the study period.
* Current active eye disease other than dry wyw syndrome (i.e., any disease for which topical or systemic ophthalmic medication is necessary).
* History of herpes keratitis.
* Corneal transplant
* Corneal refractive surgery within 6 months prior to the Screening Visit or postoperative refractive surgery symptoms of dryness that have not resolved.
* Cataract surgery within 3 months prior to the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 745 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Martel Eye Medical Group, Rancho Cordova, California
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Fifth Avenue Eye Associates, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject in OTX-101 0.09% group, was never treated with study medication and is not included in any of analysis sets Additionally, because the subjects in the ITT analysis set were analyzed as randomized, one subject who erroneously received OTX-101 0.09%, was included in the Vehicle group for purposes of efficacy analysis.
Period: Overall Study
Arm/Group | OTX-101 0.09% | Vehicle
Started | 372 | 373
Completed | 347 | 361
Not Completed | 25 | 12

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | OTX-101 0.09% | Vehicle | Total
Number analyzed (Participants) | 371 | 373 | 744
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (14.10) | 59.5 (14.68) | 59.0 (14.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 315 | 311 | 626
  Male | 56 | 62 | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 11 | 12 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 41 | 45 | 86
  White | 310 | 305 | 615
  More than one race | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Tear Production
Description: Percentage of Eyes with Increase from Baseline of ≥ 10 mm in Schirmer's Test Score
Time Frame: Baseline and 12 weeks
Population: Intent to treat population
Measure: Number; unit: Percentage of eyes
Arm/Group | OTX-101 0.09% | Vehicle
Number analyzed (Participants) | 371 | 373
Percentage of eyes | 16.6 | 9.2

2. Secondary Outcome: Conjunctival Staining
Description: change from baseline in total conjunctival staining score (lissamine green, modified National Eye Institute scale) at 12 weeks.
  Conjunctival Lissamine Green Staining Grades ranged from 0 (No punctate stain in zone) to 3 (Densely concentrated micropunctate stain spots)
Time Frame: Baseline and 12 weeks
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTX-101 0.09% | Vehicle
Number analyzed (Participants) | 371 | 373
score on a scale | -1.53 (1.927) | -1.16 (2.2064)

3. Secondary Outcome: Central Corneal Staining
Description: change from baseline in central corneal staining score (fluorescein, modified NEI/FDA scale) at 12 weeks.
  The Expanded National Eye Institute (NEI)/Industry Workshop Scale for Corneal Staining Score was used to grade each of the 5 areas of the cornea on a 0 (No punctate stain in area) to 4 (Severe diffuse (coalescent) macropunctate stain of the area) scale.
Time Frame: Baseline and 12 weeks
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTX-101 0.09% | Vehicle
Number analyzed (Participants) | 341 | 373
score on a scale | -0.28 (0.533) | -0.26 (0.588)

4. Secondary Outcome: Symptom Score
Description: change from baseline in modified Symptom Assessment in Dry Eye (SANDE) score at 12 weeks.
  A modified SANDE instrument was used to evaluate dry eye symptoms at each visit.
  Subjects were asked to indicate:
  1. frequency of dry and irritated eyes on a scale of 0 (rarely) to 100 (all the time); and
  2. severity of dry eyes on a scale of 0 (very mild) to 100 (severe) The global symptom score is the square root of the frequency score times the severity score and will be completed at each visit. (range 0 to 100)
  Negative change from baseline indicates improvement.
Time Frame: Baseline and 12 weeks
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OTX-101 0.09% | Vehicle
Number analyzed (Participants) | 371 | 373
score on a scale | -18.8 (24.08) | -19.1 (23.14)

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- OTX-101 0.09%: 0.09% cyclosporine nanomicellar ophthalmic solution.
  A total of 744 subjects were included in the Safety population, with 372 subjects in the OTX-101 0.09% group and 372 subjects in the Vehicle group. The only difference between the ITT and the Safety populations is that Subject 14-003 was analyzed in the Safety population according to the treatment received, which was OTX-101 0.09%
- Vehicle: vehicle of OTX-101
  A total of 744 subjects were included in the Safety population, with 372 subjects in the OTX-101 0.09% group and 372 subjects in the Vehicle group. The only difference between the ITT and the Safety populations is that Subject 14-003 was analyzed in the Safety population according to the treatment received, which was OTX-101 0.09%
Arm/Group | OTX-101 0.09% | Vehicle
All-Cause Mortality (participants affected / at risk) | 1/372 | 0/372
Serious Adverse Events (participants affected / at risk) | 6/372 | 2/372
Other Adverse Events (participants affected / at risk) | 130/372 | 66/372
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTX-101 0.09% (N=372) | Vehicle (N=372)
Death (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Perforated ulcer (General disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OTX-101 0.09% (N=372) | Vehicle (N=372)
Conjunctival hyperaemia (Eye disorders) | 30 | 18
Blepharitis (Eye disorders) | 5 | 0
Eye irritation (Eye disorders) | 3 | 5
Eye pruritus (Eye disorders) | 1 | 5
Instillation site pain (General disorders) | 90 | 16
Instillation site lacrimation (General disorders) | 4 | 0
Instillation site reaction (Eye disorders) | 4 | 2
Sinusitis (Eye disorders) | 4 | 5
Urinary tract infection (Eye disorders) | 4 | 2
Headache (Nervous system disorders) | 6 | 2
Foreign body sensation in eyes (Eye disorders) | 1 | 5
Conjunctival haemorrhage (Eye disorders) | 2 | 1
Posterior capsule opacification (Eye disorders) | 2 | 2
Punctate keratitis (Eye disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes